CLINICAL TRIAL: NCT05815576
Title: Lower Limb (Patho-)Mechanical Joint Contact Forces and Intrinsic Foot Muscle Properties in Subjects With Lateral Ankle Sprain and Chronic Ankle Instability
Brief Title: Biomechanics and Intrinsic Foot Muscle Roles in Subjects With Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Collaborators: UZ Leuven, campus Pellenberg (Belgium) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Screening
Other Study IDs: B3222022000964; S66498 (Other: UZ Leuven, KU Leuven, Belgium)
Record Dates: First submitted 2023-01-23; First posted 2023-04-18 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Chronic Ankle Instability; Lateral Ankle Sprain
Keywords: Biomechanical phenomena; Kinetics; Kinematics; Intrinsic foot muscles; CAI; Plantar pressures; Ultrasound

STUDY DESIGN:
Intervention Model Description: The intervention is a fatigue protocol of the intrinsic foot muscles. Only subjects with chronic ankle instability will undergo this fatigue protocol.
  Participants with chronic ankle instability will perform the movement analysis first without and then with foot muscle fatigue.
Who Masked: Outcomes Assessor
Masking Description: The data will be coded (pseudonymization). The subject's name or other identifiers will be stored separately from their research data and replaced with a unique code to create a new identity for the subject.
  The outcomes assessor will be blind for participants' injury status for the following :
  * while conducting kinematic and kinetic data processing,
  * while performing muscle size measurements on the ultrasound images,
  * while performing statistical analysis (for all outcomes)
  There will be no blinding while scoring the following outcomes (because these scores are immediately determined in the presence of the participant) :
  * Foot muscle strength,
  * Foot posture index,
  * Navicular drop,
  * Modified Star Excursion Balance Test,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intrinsic foot muscle fatigue (Experimental): The fatigue protocol will consist of repeated movements of doming (short foot exercise), combined with electrostimulation of the abductor hallucis muscle, while standing on both feet. Participants will be familiarized with doming and electrostimulation during five minutes. They will then have a rest period of at least 5 minutes The electrostimulation electrodes will be placed behind the head of the first metatarsal bone and in front of the medial tubercule of the calcaneus, on the most affected side of subjects with chronic ankle instability (according to CAIT questionnaire scores).
  Interventions: Behavioral: Intrinsic foot muscle fatigue
- No intrinsic foot muscle fatigue (No Intervention): No fatigue of the intrinsic foot muscles.

INTERVENTIONS:
Behavioral: Intrinsic foot muscle fatigue — Electrostimulation will be delivered through electrodes placed on the abductor hallucis (NOT invasive).
  The investigators plan 4 sets of 4 minutes of repeated contractions (electrostimulation + voluntary contraction).
  Arms: Intrinsic foot muscle fatigue

SUMMARY:
The current study involves a prospective interventional study that primarily intends to compare foot joint loadings of participants with chronic ankle instability (CAI) with those of subjects who recovered after an ankle sprain (LAS copers) and healthy controls during running and more challenging tasks. This study further aims to explore the impact of foot muscle properties and fatigue on the same biomechanical outcomes. Therefore, the investigators will recruit 72 participants (24 per group) aged from 18 to 44 years. Each of them will come only once to the CMAL laboratory (UZ Leuven, Pellenberg).

ELIGIBILITY:
Three groups of participants : Chronic ankle instability, lateral ankle sprain copers and healthy controls.

INCLUSION CRITERIA:

1. For all three groups :

   * Physically active male subjects between 18 and 44 years of age
   * Able to run at low speed.
   * For homogeneity purposes, the investigators will only recruit subjects who perform a regular physical activity on a weekly basis, including competition participation.
2. Chronic ankle instability :

   * A history of at least one significant ankle sprain that occurred at least 12 months before study enrolment, associated with inflammatory symptoms, creating at least 1 interrupted day of desired physical activity;
   * The most recent injury occurred more than 3 months prior to study enrolment;
   * At least two episodes of giving way in the 6 months prior to study enrolment, recurrent sprain, and/or "feelings of instability"; and
   * Poor disability status according to the Cumberland Ankle Instability Tool (CAIT) (score ≤ 24/30).
3. Lateral ankle sprain copers :

   * A history of one significant ankle sprain that occurred at least 12 months before study enrolment, associated with inflammatory symptoms, creating at least 1 interrupted day of desired physical activity;
   * A return to at least moderate levels of weight-bearing physical activity less than 12 months after initial sprain without recurrent injury, episodes of giving way, and/or feelings of instability;
   * Minimal, if any, level of self-reported disability (CAIT score ≥ 28/30); and
   * Minimal, if any, alteration in self-reported function (ADL- and Sport-subscales ≥95%).
4. Healthy controls :

   * The same inclusion criteria as the LAS coper group, with the exception reported in the exclusion criteria.

EXCLUSION CRITERIA:

1. For all three groups :

   * Being younger than 18 years
   * Any medical contraindication to physical exertion,
   * Any systemic or neurological disease,
   * A recent surgery,
   * A difference in leg length of more than 3 cm,
   * Pregnancy,
   * A body mass index higher than 30kg/m² (due to less accurate motion analysis by absence of anatomical landmarks).
   * LAS copers and controls will also be excluded if: constant or intermittent ankle pain, ankle fractures, or surgeries, and recent participation in a physical revalidation programme.
   * Healthy participants must never have suffered an inversion trauma resulting in disability.
2. For healthy controls : the healthy control subjects may not have suffered from an ankle sprain.

Ages: 18 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Lower limb joint angles | Baseline
  Part of "Kinematic data"
  Unit of measurement: Degrees
  Measurement tools: Vicon software (data acquisition) + Matlab routine (data processing)
  Method: Joint angles will be measured based on the position of passive markers placed on participants' anatomical landmarks all over the lower limbs. The position of those markers will be tracked by 10 infrared high-speed cameras that surround the walkway (sampled at 100Hz - type T-10, 1 megapixel, captures 10-bit grayscale using 1120 * 896 pixels, Vicon Motion System Ltd, Oxford, Metrics, UK).
  The angular positions of the multiple joints that constitute the lower limb (hip, knee, ankle, chopart, lisfranc and metatarsophalangeal) will be assessed during running, side-cutting and crossing over a small obstacle in the gait laboratory.
Lower limb joint angles | 5 minutes after the end of the intervention
  Part of "Kinematic data"
  Unit of measurement: Degrees
  Measurement tools: Vicon software (data acquisition) + Matlab routine (data processing)
  Method: Joint angles will be measured based on the position of passive markers placed on participants' anatomical landmarks all over the lower limbs. The position of those markers will be tracked by 10 infrared high-speed cameras that surround the walkway (sampled at 100Hz - type T-10, 1 megapixel, captures 10-bit grayscale using 1120 * 896 pixels, Vicon Motion System Ltd, Oxford, Metrics, UK).
  The angular positions of the multiple joints that constitute the lower limb (hip, knee, ankle, chopart, lisfranc and metatarsophalangeal) will be assessed during running, side-cutting and crossing over a small obstacle in the gait laboratory.
Lower limb joint angular velocities | Baseline
  Part of "Kinematic data"
  Unit of measurement: Degrees/second
  Measurement tool: Vicon software + Matlab routine
  Method: Joint angular velocities are also assessed based on reflexive markers placed on anatomical landmarks. This outcome evaluates the rate of change of a certain joint angle over time.
  Joint angular velocities will be assessed during running, side-cutting and crossing over a small obstacle in the gait laboratory.
Lower limb joint angular velocities | 5 minutes after the end of the intervention
  Part of "Kinematic data"
  Unit of measurement: Degrees/second
  Measurement tool: Vicon software + Matlab routine
  Method: Joint angular velocities are also assessed based on reflexive markers placed on anatomical landmarks. This outcome evaluates the rate of change of a certain joint angle over time.
  Joint angular velocities will be assessed during running, side-cutting and crossing over a small obstacle in the gait laboratory.
Joint moments | Baseline
  Part of "Kinetic data"
  Unit of measurement: Newton-meter
  Measurement tools: Pressure plate + Force plate + Vicon software + Matlab routine
  Methods: Joint moments will be determined by coupling kinematic data (joint position and velocities) with plantar pressure data from a specially designed pressure plate (sampled at 200Hz, Footscan, dimension 0.5m x 0.4m, 4096 sensors, 2.8 sensors/cm², RsScan International, Olen, Belgium) embedded in the middle of the runway and placed on top of a force plate (sampled at 1000Hz, Advanced Mechanical Technology Inc., Watertown, MA, USA).
  Kinetic data will be assessed while running, side-cutting and crossing over a small obstacle in the gait laboratory.
Joint moments | 5 minutes after the end of the intervention
  Part of "Kinetic data"
  Unit of measurement: Newton-meter
  Measurement tools: Pressure plate + Force plate + Vicon software + Matlab routine
  Methods: Joint moments will be determined by coupling kinematic data (joint position and velocities) with plantar pressure data from a specially designed pressure plate (sampled at 200Hz, Footscan, dimension 0.5m x 0.4m, 4096 sensors, 2.8 sensors/cm², RsScan International, Olen, Belgium) embedded in the middle of the runway and placed on top of a force plate (sampled at 1000Hz, Advanced Mechanical Technology Inc., Watertown, MA, USA).
  Kinetic data will be assessed while running, side-cutting and crossing over a small obstacle in the gait laboratory.
Joint powers | Baseline
  Part of "Kinetic data"
  Unit of measurement: Watt
  Measurement tools: Pressure plate + Vicon software + Matlab routine
  Methods: Joint moments will be determined by coupling kinematic data (joint position and velocities) with plantar pressure data from a specially designed pressure plate (sampled at 200Hz, Footscan, dimension 0.5m x 0.4m, 4096 sensors, 2.8 sensors/cm², RsScan International, Olen, Belgium) embedded in the middle of the runway and placed on top of a force plate (sampled at 1000Hz, Advanced Mechanical Technology Inc., Watertown, MA, USA).
  Kinetic data will be assessed while running, side-cutting and crossing over a small obstacle in the gait laboratory.
Joint powers | 5 minutes after the end of the intervention
  Part of "Kinetic data"
  Unit of measurement: Watt
  Measurement tools: Pressure plate + Vicon software + Matlab routine
  Methods: Joint moments will be determined by coupling kinematic data (joint position and velocities) with plantar pressure data from a specially designed pressure plate (sampled at 200Hz, Footscan, dimension 0.5m x 0.4m, 4096 sensors, 2.8 sensors/cm², RsScan International, Olen, Belgium) embedded in the middle of the runway and placed on top of a force plate (sampled at 1000Hz, Advanced Mechanical Technology Inc., Watertown, MA, USA).
  Kinetic data will be assessed while running, side-cutting and crossing over a small obstacle in the gait laboratory.
Intrinsic foot muscle thickness | Baseline
  Unit of measurement: cm
  Methods: The thickness of five intrinsic foot muscles (abductor hallucis, flexor digitorum brevis, flexor hallucis, quadratus plantae and abductor digiti minimi) will be measured on images obtained using ultrasonography.
  To obtain those images, the investigators will scan the muscles in a longitudinal view.
Intrinsic foot muscle area | Baseline
  Unit of measurement: cm² (cm square)
  Methods: The area of five intrinsic foot muscles (abductor hallucis, flexor digitorum brevis, flexor hallucis, quadratus plantae and abductor digiti minimi) will be measured on images obtained using ultrasonography.
  To obtain those images, the investigators will scan the muscles in a transversal view.

SECONDARY OUTCOMES:
Cumberland Ankle Instability Tool | Baseline
  This questionnaire assesses the level of perceived instability (higher scores indicate less self-reported instability).
  Scores ranging from 0 to 30.
  The CAIT is valid and reliable, and has known minimal detectable changes. It has been validated in French and Dutch.
  This is an inclusion questionnaire.
Foot and Ankle Activity Measure | Baseline
  This questionnaire assesses the level of self-reported functional limitations (higher scores indicate less limitations).
  Score ranging from 0 to 100%
  The FAAM is valid, reliable and responsive to change. It has been validated in French and Dutch. It contains two subscales: Activity of Daily Life (ADL) and Sports. A "Quick" version has shown strong concurrent validity with the full-length FAAM.
  This is an inclusion questionnaire
Ankle-specific Fear-Avoidance Beliefs Questionnaire | Baseline
  This questionnaire is an adapted version of the original FABQ designed to assess kinesiophobia in people with low-back pain. The term "back" was changed to "ankle" and item 8 of the original FABQ was deleted. It contains two subscales: Physical Activity and Work.
  Higher scores indicate more kinesiophobia. Scores ranging from 0 to 90.
  The ankle-specific FABQ has shown acceptable internal consistency, and its use is encouraged in people with a history of ankle sprain, with known minimal detectable change. The FABQ questionnaire was validated in French, and a non-validated Dutch version was published.
Foot muscle strength | Baseline
  Unit of measurement: Newton
  Method: Foot muscle strength will be evaluated using a hand-held dynamometer, with participants hook lying. The investigators will both report the strength of the big toe and the strength of the other toes (as a whole). This method showed good to excellent intra and inter-rater reliability.
Change from baseline in hallux flexion strength after the intervention | Change between baseline and immediately post-intervention
  Unit of measurement: Newton
  Method: Hallux flexion strength will be evaluated using a hand-held dynamometer, with participants hook lying.
  The difference between before and after the intervention (fatigue protocol) will be reported.
Foot Posture Index | Baseline
  No unit of measurement.
  The Foot Posture Index 6-item is a valid measure of foot posture (pronation, neutral and supination). Its reliability is subject of debate, ranging from poor to excellent for inter-rater and from moderate to excellent for intra-rater. The participants will stand bilaterally in a static position during the assessment.
Navicular drop | Baseline
  Unit of measurement: cm
  The investigators will assess navicular drop as the difference in distance between the navicular tuberosity to the ground from sitting to double-limb stance
Modified Star Excursion Balance Test | Baseline
  Unit of measurement: cm
  The modified Star Excursion Balance Test assesses dynamic balance. In recent studies involving subjects with CAI, the mSEBT was preferred over the original eight-direction version because the former measures are the most often altered in this population and the remaining directions add thus little value.
  The original SEBT is reliable, valid, reproducible, and responsive to change.
  The modified SEBT requires the participant to reach the ground as far as possible with his leg in the anterior, postero-medial and postero-lateral directions. The procedure is repeated until three valid trials are measured in each direction for each leg.
  A mean score will then be calculated for each direction as the mean of the three valid trials with one leg. Those values will first be normalized by the leg length and a composite score will then be calculated as the mean of the three directions reached with one leg.
Perceived foot fatigue | 4 minutes after the beginning of the intervention
  No unit of measurement.
  Participants will be asked to score their perceived foot fatigue every four minutes during the fatigue protocol.
  This will be done based on a verbal scale from 0 (no perceived fatigue at all) to 10 (highest fatigue the participant could imagine).
  The foot muscle fatigue protocol lasts 16 minutes. Time frame 16 minutes is thus equal to "immediately post-intervention".
Perceived foot fatigue | 8 minutes after the beginning of the intervention
  NB: Same as above
  No unit of measurement.
  Participants will be asked to score their perceived foot fatigue every four minutes during the fatigue protocol.
  This will be done based on a verbal scale from 0 (no perceived fatigue at all) to 10 (highest fatigue the participant could imagine).
  The foot muscle fatigue protocol lasts 16 minutes. Time frame 16 minutes is thus equal to "immediately post-intervention".
Perceived foot fatigue | 12 minutes after the beginning of the intervention
  NB: Same as above
  No unit of measurement.
  Participants will be asked to score their perceived foot fatigue every four minutes during the fatigue protocol.
  This will be done based on a verbal scale from 0 (no perceived fatigue at all) to 10 (highest fatigue the participant could imagine).
  The foot muscle fatigue protocol lasts 16 minutes. Time frame 16 minutes is thus equal to "immediately post-intervention".
Perceived foot fatigue | Immediately after the end of the intervention
  NB: Same as above
  No unit of measurement.
  Participants will be asked to score their perceived foot fatigue every four minutes during the fatigue protocol.
  This will be done based on a verbal scale from 0 (no perceived fatigue at all) to 10 (highest fatigue the participant could imagine).
  The foot muscle fatigue protocol lasts 16 minutes. Time frame 16 minutes is thus equal to "immediately post-intervention".
Electrostimulation current intensity | 4 minutes after the beginning of the intervention
  Unit of measurement: mA (milli-amperes).
  Every 4 minutes, electrostimulation current intensity will be reported during the foot muscle fatigue protocol.
  NB: This current intensity should gradually increase during the fatigue protocol as there is a habituation phenomenon. In other words, constant intensity produces decreasing discomfort.
  The foot muscle fatigue protocol lasts 16 minutes. Time frame 16 minutes is thus equal to "immediately post-intervention".
Electrostimulation current intensity | 8 minutes after the beginning of the intervention
  NB: Same as above
  Unit of measurement: mA (milli-amperes).
  Every 4 minutes, electrostimulation current intensity will be reported during the foot muscle fatigue protocol.
  NB: This current intensity should gradually increase during the fatigue protocol as there is a habituation phenomenon. In other words, constant intensity produces decreasing discomfort.
  The foot muscle fatigue protocol lasts 16 minutes. Time frame 16 minutes is thus equal to "immediately post-intervention".
Electrostimulation current intensity | 12 minutes after the beginning of the intervention
  NB: Same as above
  Unit of measurement: mA (milli-amperes).
  Every 4 minutes, electrostimulation current intensity will be reported during the foot muscle fatigue protocol.
  NB: This current intensity should gradually increase during the fatigue protocol as there is a habituation phenomenon. In other words, constant intensity produces decreasing discomfort.
  The foot muscle fatigue protocol lasts 16 minutes. Time frame 16 minutes is thus equal to "immediately post-intervention".
Electrostimulation current intensity | Immediately after the end of the intervention
  NB: Same as above
  Unit of measurement: mA (milli-amperes).
  Every 4 minutes, electrostimulation current intensity will be reported during the foot muscle fatigue protocol.
  NB: This current intensity should gradually increase during the fatigue protocol as there is a habituation phenomenon. In other words, constant intensity produces decreasing discomfort.
  The foot muscle fatigue protocol lasts 16 minutes. Time frame 16 minutes is thus equal to "immediately post-intervention".

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Deschamps, Principal Investigator — Musculoskeletal Rehabilitation Research Group, Department of Rehabilitation Sciences, KU Leuven; Christine Detrembleur, Principal Investigator — Neuro Musculo Skeletal Lab (NMSK), IREC, SSS, UCLouvain
Locations (1):
- UZ Leuven, Pellenberg, Lubbeek, Belgium

IPD SHARING:
Plan to Share IPD: No